CLINICAL TRIAL: NCT06636721
Title: Lung Cancer and Aging (LuCA): Intervention Development for Addressing Aging-specific Concerns in Older Adults With Lung Cancer
Brief Title: Lung Cancer and Aging: Improving Well-being for Older Adults With Lung Cancer
Acronym: LuCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00116551; 5T32AG000029-47 (NIH)
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
Keywords: aging; depression; anxiety; pain; dyspnea; behavioral medicine; psycho-oncology
MeSH Terms: conditions — Lung Neoplasms; Depression; Anxiety Disorders; Pain; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Intervention (Experimental): Participants will engage in a 5-session protocol, to be delivered in an individual therapy setting, via telehealth or in-person. The program will integrate aspects of Cognitive Behavioral Therapy and Acceptance and Commitment Therapy.
  Interventions: Behavioral: LuCA Behavioral Intervention

INTERVENTIONS:
Behavioral: LuCA Behavioral Intervention — The intervention will integrate aspects of Cognitive Behavioral Therapy (identifying and challenging automatic thoughts, engaging in behavioral activation) and Acceptance and Commitment Therapy (integrating one's values, distancing skills). The intervention will include skills such as problem-solving, communicating with close others and the medical team, and breathing techniques to improve shortness of breath related to lung cancer.

SUMMARY:
The purpose of this study is to develop a brief assessment and need-based behavioral intervention for addressing aging-specific concerns in older adults with lung cancer. The long-term goals of this research include identifying the unique concerns of these patients, providing patients with behavioral skills to address their symptom management needs, and enhancing patient engagement with healthcare specialties targeting aging-specific concerns.

In the first phase of this study, participants (12 patients with lung cancer, 6 caregivers, 12 providers) will be asked to participate in two individual interviews (each 30-45 minutes in length) via teleconference. During the first interview, participants will be asked to provide feedback on the current version of the assessment and behavioral intervention. Participants will be asked to describe strengths and weaknesses of the materials, topics to add or remove, and any other suggested changes. After the research team has made changes to the materials, participants will be invited to complete a second interview to provide feedback on the updated materials.

In the second phase of the study, 16 older adults with lung cancer will complete the revised assessment and participate in the behavioral intervention, in order to a) evaluate the feasibility and acceptability of the program and b) measure change in depression, anxiety, pain, and dyspnea.

DETAILED DESCRIPTION:
Aim 1. The investigators will first develop a brief geriatric assessment, designed to address the specific needs of older adults with lung cancer. As a foundation, the investigators will collect existing, empirically supported geriatric assessment tools, such as the Senior Adult Oncology Program (SAOP) assessment and the Geriatric 8 (G8), and the Triage Risk Screening Tool (TRST). The investigators will combine these tools such that all relevant domains are included in the aggregated assessment. The study team will then collaboratively add further items into the assessment (as related to difficulties commonly faced by older adults with lung cancer) and remove excess or irrelevant items.

The study team will then develop the initial prototype of a need-based behavioral intervention protocol to address aging-specific concerns and multimorbidity in older adults with lung cancer. The behavioral intervention will build upon and extend a previously tested intervention, which demonstrated benefits for reducing depressive and anxiety symptoms in older adults with lung cancer. The intervention will be a 5-session protocol, to be delivered to patients in an individual therapy setting, via telehealth or in-person. The program will integrate aspects of cognitive behavioral therapy (identifying and challenging automatic thoughts, engaging in behavioral activation) and acceptance and commitment therapy (integrating one's values, distancing skills). The intervention will include skills such as problem-solving, communicating with close others and the medical team, and breathing techniques to improve shortness of breath related to lung cancer.

Aim 2. The investigators will then conduct interviews with lung cancer patients (N=12), provider stakeholders (N=12), and caregivers (N=6) in order to obtain feedback on the proposed assessment and intervention. Caregiver participants will be either a) caregivers for lung cancer patients participating in interviews for this study, or b) caregivers for other patients with lung cancer. Each interview will be 30-45 minutes in length.

All patient, caregiver, and provider interview sessions will be recorded and transcribed verbatim. During interview sessions, the participant will be provided with the current version of the geriatric assessment and behavioral intervention. A semi-structured interview script will be utilized to obtain feedback on the strengths and weaknesses of the materials, thoughts on topics to add or remove, and amendments to any wording or structural details. Data from the initial interviews will allow the investigators to refine the assessment, referral resources, and intervention content so that it best meets the needs of this patient population.

All patients, caregivers, and provider stakeholders will be invited to complete a second interview to provide feedback on the revised materials. Thus, participants will be recruited to participate in 2 interviews - one for the initial set of materials, and one for the revised set. Because all participation is voluntary, participants can choose to opt out of any portion. If the investigators are unable to obtain adequate response rates for the second interview, they will recruit new participants meeting eligibility criteria to complete interviews surrounding the revised material.

Aim 3. The investigators will then conduct a preliminary study to evaluate the feasibility and acceptability of the revised geriatric assessment and behavioral intervention protocol. N=16 older adults with lung cancer will be recruited to complete the geriatric assessment and 5-session intervention. The assessment will be completed on paper in the clinic or digitally via RedCap survey sent via email, based on participant preference. The intervention sessions will be conducted via telehealth. Sessions will occur once per week for 5 weeks, and will last approximately one hour each. Sessions will be video-recorded and transcribed verbatim.

ELIGIBILITY:
Inclusion Criteria for Patient Participants:

* Lung cancer diagnosis
* 60 years of age or older
* Receiving active treatment at Duke University Health System
* Able to speak/read English and provide informed consent

Inclusion Criteria for Caregiver Participants:

* Caregiver for a patient with lung cancer participating in this study
* Caregiver for other patient with lung cancer
* Able to speak/read English and provide informed consent

Inclusion Criteria for Provider Participants:

* Provide care for older adults with lung cancer
* Able to speak/read English and provide informed consent

Exclusion Criteria for all:

* Visual or hearing impairment, cognitive impairment, or severe mental illness interfering with participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by number of recruited participants who enrolled | 5 weeks
  Study feasibility will be measured by number of recruited participants who enroll.
Feasibility as measured by number of participants who completed all study activities | 5 weeks
  Feasibility of the study will be measured by number of participants who complete all study activities.
Acceptability as measured by Study Satisfaction Questionnaire | 5 weeks
  Acceptability of the study will be measured by the Study Satisfaction Questionnaire. This is a 15-item measure using a 5-point Likert scale (from "strongly disagree" to "strongly agree") in which a higher score indicates greater satisfaction.

SECONDARY OUTCOMES:
Change in depressive symptoms as measured by the Patient Health Questionnaire (PHQ-9) | Baseline to 5 weeks
  The Patient Health Questionnaire-9 total score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression).
Change in anxiety symptoms as measured by the Generalized Anxiety Disorder (GAD-7) scale | Baseline to 5 weeks
  The Generalized Anxiety Disorder-7 score ranges from 0 to 21, where a higher score indicates greater anxiety.
Change in physical pain as measured by the Brief Pain Questionnaire (BPI) | Baseline to 5 weeks
  The Brief Pain Inventory (BPI) is a tool that uses a numeric rating scale (NRS) from 0 to 10, where a higher score indicates greater pain.
Change in dyspnea as measured by the Chronic Respiratory Questionnaire (CRQ) | Baseline to 5 weeks
  The Chronic Respiratory Questionnaire is scored on a 7-point scale, with 1 indicating maximum impairment and 7 indicating no impairment. Higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Shelby, PhD, Principal Investigator — Duke Psychiatry & Behavioral Sciences
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
It is the investigators' intention to make all data generated from this study freely available after it is de-identified. All direct respondent identifiers (e.g., names and addresses) will be removed and maintained in a secure file for future contact purposes. Respondent identifiers will not be shared. All other scientific data (scale composites) will be both preserved and shared. The following data will be preserved and shared: patient-reported data from study assessments, assessment and intervention utilization data, healthcare utilization data collected from the health record, and socio-demographic and medical data collected via patient report and health record. The investigators will make every effort to provide raw data in a non-proprietary format wherever possible to enhance reproducibility.